CLINICAL TRIAL: NCT04177563
Title: Impact of Systemic Cryotherapy on the Rheological, Morphological, and Biochemical Blood Indicators
Brief Title: Whole Body Cryotherapy and Morphological and Rheological Indicators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University School of Physical Education, Krakow, Poland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: USPKrakow
Record Dates: First submitted 2019-11-13; First posted 2019-11-26 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2014-11

CONDITIONS: Quality of Life
Keywords: whole-body cryotherapy; healthy men; blood components

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- a group of ten students with high physical activity (Experimental): The participants of the study were subjected to 24 whole-body cryotherapy treatments (one treatment three times a week for two months). Before the procedure, they were informed about how to move and breathe in the cryochamber. Each entrance to the cryochamber was preceded by a 30-second adaptation period in the vestibule at a temperature of -60 ºC. Then the subjects entered the cryochamber for three minutes.
  Blood was collected from each participant (with an empty stomach) at a laboratory located at the Academy of Physical Education in Krakow, where after a ten-minute rest in a sitting position at room temperature (about 19 °C), blood was collected from the vein in the crook of the elbow by a laboratory diagnostician in accordance with applicable standards. Blood was collected 13 times.
  Interventions: Other: whole body cryostimulation
- a group of eight students with moderate physical activity (Experimental): The participants of the study were subjected to 24 whole-body cryotherapy treatments (one treatment three times a week for two months). Before the procedure, they were informed about how to move and breathe in the cryochamber. Each entrance to the cryochamber was preceded by a 30-second adaptation period in the vestibule at a temperature of -60 ºC. Then the subjects entered the cryochamber for three minutes.
  Blood was collected from each participant (with an empty stomach) at a laboratory located at the Academy of Physical Education in Krakow, where after a ten-minute rest in a sitting position at room temperature (about 19 °C), blood was collected from the vein in the crook of the elbow by a laboratory diagnostician in accordance with applicable standards. Blood was collected 13 times.
  Interventions: Other: whole body cryostimulation

INTERVENTIONS:
Other: whole body cryostimulation — Whole-body cryotherapy

SUMMARY:
The aim of the planned study was to evaluate the effect of repeated cryostimulation treatments on immunological, morphological, and biochemical indicators of the peripheral blood of healthy, young Men

DETAILED DESCRIPTION:
A group of 18 healthy men aged 19-26 participated in the study. The group included a group of ten students with high physical activity and a group of eight students with moderate physical activity.

Whole-body cryotherapy was performed in a cryochamber located in the Malopolska Cryotherapy Centre in Krakow (Poland) in the spring of 2013 and in the winter and spring of 2014.

The temperature inside the vestibule during the procedure was about -60 ºC and in the actual chamber about -120 ºC. The concentration of oxygen in the air of the cryochamber was kept constant at 21-22% and continuously controlled by two independent oxygen probes.

The participants of the study were subjected to 24 whole-body cryotherapy treatments (one treatment three times a week for two months). Before the procedure, they were informed about how to move and breathe in the cryochamber. Each entrance to the cryochamber was preceded by a 30-second adaptation period in the vestibule at a temperature of -60 ºC. Then the subjects entered the cryochamber for three minutes. During the treatment, the men wore short trousers, woollen socks and gloves, hats or headbands to protect against freezing and clogs. Moreover, the mouths and noses of the participants were covered with surgical masks, secured with a strip of gauze. During the procedure, the subjects were in permanent eye contact with the doctor and the staff.

ELIGIBILITY:
Inclusion Criteria:

* informed consent for research;
* equal age and above 18 years of age;
* no contraindications to cryostimulation procedures;
* physically active

Exclusion Criteria:

* lack of informed consent for research
* children and adolescents under 18 years of age,
* patients with inflammatory diseases, infectious, autoimmune and cancer

Ages: 18 Years to 27 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2015-12-20 (Actual); Study Completion 2015-12-20 (Actual)

PRIMARY OUTCOMES:
blood collection in a group of participants with high and moderate physical activity | up to 3 months
  Determination of blood components

SECONDARY OUTCOMES:
blood collection in both groups tested | for 3 months
  Determination of blood rheology

OTHER OUTCOMES:
Research in both groups | through study completion, an average of 1 month
  determination of blood biochemical components

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Kepinska-Szyszkowska, PhD, Principal Investigator — University of Physical Education in Krakow, Poland

IPD SHARING:
Plan to Share IPD: No